CLINICAL TRIAL: NCT00647127
Title: Investigation of Analgesic and Anti-hyperalgesic Effect of Opioids in Experimental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2007-004524-21
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Pain
Keywords: Buprenorphine; Fentanyl; Analgesic effect; Anti-hyperalgesic effect; Experimental pain
MeSH Terms: conditions — Pain | interventions — Buprenorphine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Buprenorphine (Active Comparator)
  Interventions: Drug: Buprenorphine
- Fentanyl (Active Comparator)
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine: 20microg/h
  Other Names: Norspan
  Arms: Buprenorphine
Drug: Fentanyl — Fentanyl: 25microg/h
  Other Names: Durogesic
  Arms: Fentanyl
Drug: Placebo — Placebo: '5microg/h' (not active drug, it is just called '5microg/h')
  Other Names: Norspan
  Arms: Placebo

SUMMARY:
To compare the analgesic and anti-hyperalgesic effect of Buprenorphine and Fentanyl against experimental pain in skin, muscle and bone. The study will be performed with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* men > 18 years

Exclusion Criteria:

* women
* known allergy against the investigated drugs
* ongoing participation in other experiments or participation in other experiments 14 days before screening
* previously pain or psychiatric conditions
* simultaneously use of pain killers
* alcohol
* previously drug-addict or member of family with drug-addicts
* chronic constipation
* ileus
* inflammatory bowel syndrome
* abdominal surgery within the last three months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Data will be electronically recorded or written directly in case report form. Outcome measure will be a subjective rating of the pain with a visual analogue scale. | Continuously

CONTACTS AND LOCATIONS:
Overall Officials: Asbjoern M Drewes, MD, Prof., Principal Investigator — Mech Sense, Department of Gastroenterology, Aalborg Hospital
Locations (1):
- Mech Sense, Department of Gastroenterology, Aalborg, Region Nordjyllan, Denmark